CLINICAL TRIAL: NCT02350881
Title: A Post-Market Observational Study to Evaluate Safety and Performance of Primus™ FGT Implant at a Minimum of 5 Years Follow-up
Brief Title: Mid-term Outcomes of First MTP Arthroplasty With Primus™ FGT Implant.
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 1202-T-FGTI-M
Record Dates: First submitted 2015-01-19; First posted 2015-01-30 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-05

CONDITIONS: Hallux Limitus of Left Great Toe; Rheumatoid Arthritis; Arthritis of 1st Metatarsophalangeal Joint; Osteoarthritis; Bunion; Hallux Limitus of Right Great Toe
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Bunion

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Primus FGTI (Flexible Great toe Implant) — Great toe arthroplasty consists of replacing the first Meta-Tarso-Phalangeal (MTP1) joint by a two hinged prosthesis made of silicone : the Primus FGT implant (FGTI). The Primus is designed with an axially offset hinge to align with the anatomy of the MTP joint. This results in less implant stresses and improved toe function.
  Other Names: First metatarsophalangeal arthroplasty

SUMMARY:
Foot silicone implants suffer from bad reputation on the market, due to poor results obtained with the first generations of implants. Allergies to silicone, infections due to silicone and implants breakage used to be common with previous generations of silicone implants. Publications relative to those implants showed that the survival rates after 5 years of follow-up were unsatisfactory.

Since 1998, Tornier has been selling a new generation of silicone implants made of Ultrasil™. The use of this new material in its manufacturing process together with its innovative geometry, make the Primus™ FGT a much more resistant, anatomic and long lasting implant.

The main objective of this study is to evaluate the clinical outcomes of the implantation of Primus™ FGT implant in great toe arthroplasty. The study will capture long term outcomes in terms of functional metrics from documented clinical data. Other objectives are to evaluate the outcomes in terms of radiological evaluation and of safety during all the follow-up.

DETAILED DESCRIPTION:
This is an observational post-marketing surveillance study, performed by 1 (one) investigator in 1 (one) Italian site.

* Preoperative and peroperative data were collected retrospectively.
* Postoperative data (minimum 5 years follow-up or until implant revision) were collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* patient has had a Primus™ FGT implantation for one of the following indications: hallux limitus, hallux rigidus, hallux abducto valgus associated with severe arthritis, unstable or painful joint from previous surgery on the great toe,
* patient having all necessary clinical and radiographical data available.,
* patient has been informed about this scientific study and has provided their Consent to participate.

Exclusion Criteria:

* patient does not have clinical and radiographic follow-up data available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study has included all patients who had had a Primus™ FGT implantation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano FIESCHI, MD, Principal Investigator — Casa di Cura Villa Berica - Vicenza - Italy
Locations (1):
- Casa Di Cura Villa Berica, Vicenza, Vicenza, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period : from September 2013 to April 2014
Groups:
- Overall Cohort: one consecutive series of patients were included
Period: Overall Study
Arm/Group | Overall Cohort
Started | 64 (64 patients were included (6 bilateral))
Completed | 64 (64 patients were completed (6 bilateral))
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 64 patients who received 70 implants (6 bilateral)
Arm/Group | Overall Cohort
Number analyzed (Participants) | 64
Age, Continuous [Mean (Full Range); unit: years] | 59.8 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 18
Region of Enrollment [Number; unit: participants]
  Italy | 64

OUTCOME MEASURES:

1. Primary Outcome: AOFAS Hallux-MTP-IP Score - Overall
Description: AOFAS (American Orthopedic Foot and Ankle Society) Hallux-MTP-IP (Hallux-Meta-Tarso-Phalangeal-Inter-Phalangeal) score is composed of 3 sub-scores : (i) Pain score is ranging from 0 to 40 points ; Function score is ranging from 0 to 45 points ; Alignment is ranging from 0 to 15 points. The AOFAS total score is then ranging from 0 to 100 points. A result over 80 points is considered "good", below 20 points as "bad".
Time Frame: mean 6.9 years follow-up (range 5.2 - 9.5)
Population: number of implants analyzed (70 implants in 64 patients)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of Implants
Arm/Group | Overall Cohort
Number analyzed (Participants) | 64
Number analyzed (Number of Implants) | 70
units on a scale | 88.9 (9.1)

2. Primary Outcome: AOFAS Hallux-MTP-IP - PAIN Score
Description: Pain is a sub-score of the AOFAS Hallux-MTP-IP score and is measured on a scale of 40 points - the higher value represents a minimal pain.
Time Frame: mean follow-up of 6.9 years (range, 5.2 - 9.5)
Population: Overall cohort
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number of Implants
Arm/Group | Overall Cohort
Number analyzed (Participants) | 64
Number analyzed (Number of Implants) | 70
units on a scale | 35.4 (5.0)

3. Primary Outcome: Pain at Passive Motion of MTP1
Description: Number of patients reporting pain at passive motion of MTP1 at preoperative and postoperative visits.
Time Frame: mean follow-up of 6.9 years (range, 5.2 - 9.5)
Population: Overall cohort
Measure: Number; unit: Number of Implants
Units Other Than Participants: Number of Implants
Groups:
- Absent: Number of patients reporting no pain
- Moderate: Number of patients reporting a moderate pain
- Severe: Number of patients reporting a severe pain
Arm/Group | Absent | Moderate | Severe
Number analyzed (Participants) | 64 | 64 | 64
Number analyzed (Number of Implants) | 70 | 70 | 70
Number of Implants
  Preoperative | 0 | 6 | 64
  Postoperative | 65 | 3 | 2

4. Secondary Outcome: Osteolysis
Description: Osteolysis evaluation was described as : absent or present. Radiological evaluations were done from available frontal and lateral view X-rays.
Time Frame: mean 6.9 years (range, 5.5 - 9.5)
Population: Overall cohort
Measure: Number; unit: percentage of implants
Units Other Than Participants: Number of Implants
Groups:
- Absence: Number of feet where no osteolysis was observed
- Presence: Number of feet where osteolysis was observed
Arm/Group | Absence | Presence
Number analyzed (Participants) | 64 | 64
Number analyzed (Number of Implants) | 70 | 70
percentage of implants | 81.4 | 18.6

5. Secondary Outcome: Bone Resorption
Description: Bone resorption evaluation was described as : absent or present. Radiological evaluations were performed from available frontal and lateral view X-rays.
Time Frame: mean 6.9 years (range, 5.5 - 9.5)
Population: Overall cohort
Measure: Number; unit: percentage of implants
Units Other Than Participants: Number of Implants
Groups:
- Absence: Number of feet where no bone resorption was observed
- Presence: Number of feet where bone resorption was observed
Arm/Group | Absence | Presence
Number analyzed (Participants) | 64 | 64
Number analyzed (Number of Implants) | 70 | 70
percentage of implants | 64.3 | 35.7

6. Primary Outcome: Pain at Pressure of MTP1
Description: Number of patients reporting pain at pressure of MTP1 at preoperative and postoperative visits.
Time Frame: mean follow-up of 6.9 years (range, 5.2 - 9.5)
Population: Overall cohort
Measure: Number; unit: Number of Implants
Units Other Than Participants: Number of Implants
Groups:
- Moderate: umber of patients reporting a moderate pain
Arm/Group | Absent | Moderate | Severe
Number analyzed (Participants) | 64 | 64 | 64
Number analyzed (Number of Implants) | 70 | 70 | 70
Number of Implants
  Preperative | 0 | 16 | 54
  Postoperative | 61 | 8 | 1

7. Primary Outcome: Walking Perimeter
Description: Subjective evaluation by the patients of their walking perimeter, postoperatively versus preoperatively. Patient had to choose among 3 variables : "improved", "same", "worsened".
Time Frame: mean follow-up of 6.9 years (range, 5.2 - 9.5)
Population: Overall cohort
Measure: Number; unit: Number of Implants
Units Other Than Participants: Number of Implants
Groups:
- Improved: Number of patients who declared an improvement in their walking perimeter
- Same: Number of patients who declared no improvement in their walking perimeter
- Worsened: Number of patients who declared a worsening of their walking perimeter
Arm/Group | Improved | Same | Worsened
Number analyzed (Participants) | 64 | 64 | 64
Number analyzed (Number of Implants) | 70 | 70 | 70
Number of Implants | 59 | 11 | 0

8. Primary Outcome: Pain During Walking
Description: Subjective evaluation by patients about pain during walking, postoperatively versus preoperatively. Patients had to choose among 4 variables : "disappeared", "less", same", "greater".
Time Frame: mean follow-up of 6.9 years (range, 5.2 - 9.5)
Population: Overall cohort
Measure: Number; unit: Number of Implants
Units Other Than Participants: Number of Implants
Groups:
- Disappeared: Number of patients who declared an absence of pain during walking postoperatively
- Less: Number of patients who declared a slight improvement of pain during walking postoperatively
- Same: Number of patients who declared no improvement in pain during walking postoperatively
- Greater: Number of patients who declared a worsening of pain during walking postoperatively
Arm/Group | Disappeared | Less | Same | Greater
Number analyzed (Participants) | 64 | 64 | 64 | 64
Number analyzed (Number of Implants) | 70 | 70 | 70 | 70
Number of Implants | 55 | 15 | 0 | 0

9. Primary Outcome: Pain at Rest
Description: Subjective evaluation of patients about ther pain at rest, postoperatively versus preoperatively. Patients had to choose among 4 variables : "disappeared", "less", "same, "greater".
Time Frame: mean follow-up of 6.9 years (range, 5.2 - 9.5)
Population: Overall cohort
Measure: Number; unit: Number of Implants
Units Other Than Participants: Number of Implants
Groups:
- Disappeared: Number of patients who declared an absence of pain at rest postoperatively
- Less: Number of patients who declared a slight improvement of pain at rest postoperatively
- Same: Number of patients who declared no improvement in pain at rest postoperatively
- Greater: Number of patients who declared a worsening of pain at rest postoperatively
Arm/Group | Disappeared | Less | Same | Greater
Number analyzed (Participants) | 64 | 64 | 64 | 64
Number analyzed (Number of Implants) | 70 | 70 | 70 | 70
Number of Implants | 61 | 9 | 0 | 0

10. Secondary Outcome: Survival of the Implant.
Description: The survival of the implant is evaluated according to the number of implant revisions or of reoperations, whatever the reason.
Time Frame: mean follow-up of 6.9 years (range, 5.2 - 9.5)
Population: Overall cohort
Measure: Number; unit: percentage of implants
Units Other Than Participants: Number of Implants
Groups:
- Survival: Percentage of feet with implant still in place
- Revisions: Percentage of feet reoperated for implant ablation
Arm/Group | Survival | Revisions
Number analyzed (Participants) | 64 | 64
Number analyzed (Number of Implants) | 70 | 70
percentage of implants | 100 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the longest study follow-up, i.e. 144 months.
Arm/Group | Overall Cohort
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 1/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Cohort (N=64)
superficial skin infection around the wound (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
* inclusion of patients from only 1 site, operated by a single surgeon
* lack of control group for comparison with another treatment option
* inability to compare preoperative and postoperative AOFAS scores

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No